CLINICAL TRIAL: NCT00209261
Title: A 6-week Open Label Cross-over Study With 2 Different Daily Doses of Minirin® Oral Lyophilisate (120 μg and 240 μg) and 2 Different Daily Doses of Minirin® Tablet (0.2 mg and 2 x 0.2 mg) in Children and Adolescents With Primary Nocturnal Enuresis (PNE)
Brief Title: A 6-week Open Label Cross-over Study With 2 Different Daily Doses of Minirin® Oral Lyophilisate in Children and Adolescents With Primary Nocturnal Enuresis (PNE)
Acronym: PALAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FE992026 CS022
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Primary Nocturnal Enuresis
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: MINIRIN Oral Lyophilisate
- 2 (Active Comparator)
  Interventions: Drug: Minirin tablet

INTERVENTIONS:
Drug: MINIRIN Oral Lyophilisate
  Arms: 1
Drug: Minirin tablet
  Arms: 2

SUMMARY:
To evaluate the preference of subjects for Minirin® oral lyophilisate treatment compared with Minirin® tablet treatment after 6 weeks.

To compare efficacy of the 2 formulations at the end of the 6-week treatment period using diary card data.

To compare ease of use of both formulations at 3 and 6 weeks using a VAS-scale. To validate a PNE Quality of Life (QoL) questionnaire. To evaluate safety. To compare compliance with the 2 formulations

DETAILED DESCRIPTION:
To evaluate the preference of subjects for Minirin® oral lyophilisate treatment compared with Minirin® tablet treatment after 6 weeks.

To compare efficacy of the 2 formulations at the end of the 6-week treatment period using diary card data.

To compare ease of use of both formulations at 3 and 6 weeks using a VAS-scale. To validate a PNE Quality of Life (QoL) questionnaire. To evaluate safety. To compare compliance with the 2 formulations

ELIGIBILITY:
Inclusion Criteria:

* Children suffering from primary nocturnal enuresis with no organic pathology.
* Children of either sex, not below 5 and not above 15 years of age (not below 6 years in The Netherlands and France).
* Children with a minimum of 6 wet nights in 2 weeks.

Exclusion Criteria:

* Children who have previously been treated with desmopressin or other medications for nocturnal enuresis or enuresis alarms.
* Children receiving substances that are known or suspected to potentiate antidiuretic hormone, e.g. SSRI, tricyclic antidepressant drugs, chlorpromazine and carbamazepine.
* Diagnosed renal diabetes insipidus or central diabetes insipidus with an AVP (arginine vasopressin) deficiency.
* Proven urinary tract infection within the past month or a documented positive urine culture at the start of the study

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2004-12; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the difference in the proportion of subjects who preferred each formulation at the end of the 6-week treatment period. | 6 weeks (melt) and 6 weeks (tablet). Total 12 weeks.

SECONDARY OUTCOMES:
Efficacy will be measured as the difference in the incidence of bedwetting episodes during each 3-week treatment period, compared between formulations. | 3 weeks
The subjects will be asked to rate the ease of use of each formulation using a 100 mm Visual Analogue Scale (VAS), with 0 = I find it very easy to use this medicine and 100 = I find it very difficult to use this medicine. | 3 weeks
Subjects will be asked to complete a QoL questionnaire at visit 2 and visit 3. | 3 weeks
Safety comparison between the 2 formulations. | 6 weeks
Comparison of compliance between the 2 formulations. | 6 weeks
The subjects will be asked a question regarding which treatment (Minirin® oral lyophilisate or Minirin® tablet) they preferred at the end of 6 weeks treatment. | 6 weeks (melt) and 6 weeks (tablet). Total 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Service de Chirurrgie Viscerale Pediatrique Hospital Necker-Enfants Malades, Paris, France

REFERENCES:
- [Derived] Hahn D, Stewart F, Raman G. Desmopressin for nocturnal enuresis in children. Cochrane Database Syst Rev. 2025 Jul 29;7(7):CD002112. doi: 10.1002/14651858.CD002112.pub2. PMID 40728007
- [Derived] Caldwell PH, Codarini M, Stewart F, Hahn D, Sureshkumar P. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2020 May 4;5(5):CD002911. doi: 10.1002/14651858.CD002911.pub3. PMID 32364251
- [Derived] Juul KV, Van Herzeele C, De Bruyne P, Goble S, Walle JV, Norgaard JP. Desmopressin melt improves response and compliance compared with tablet in treatment of primary monosymptomatic nocturnal enuresis. Eur J Pediatr. 2013 Sep;172(9):1235-42. doi: 10.1007/s00431-013-1992-9. Epub 2013 May 16. PMID 23677249